

# Non-Interventional Study C4671054

A Retrospective Observational Non-Interventional Study (NIS) to assess Patient Characteristics and Healthcare Resource Use (HCRU) among COVID-19 Patients Receiving Treatment with Nirmatrelvir; Ritonavir (PAXLOVID TM) in the Kingdom of Saudi Arabia (KSA)

Statistical Analysis Plan (SAP)

Version: 2

Author: PPD

(PPC

IQVIA)

Date: 16th September 2024

# **TABLE OF CONTENTS**

| 1 | LIS | T OF ABBREVIATIONS | 3 |
|---|---|---|---|
| 2 | AM | ENDMENTS FROM PREVIOUS VERSION(S) | 5 |
| 3 | INT | RODUCTION | 7 |
| | 3.1<br>3.1.<br>3.1.<br>3.1.<br>3.1.<br>3.2<br>3.2.<br>3.2. | 2 Inclusion Criteria | 11 12 12 12 13 13 |
| 4 | AN | ALYSIS SETS/POPULATIONS | 14 |
| | 4.1<br>4.2 | FULL ANALYSIS SET | |
| 5 | ENI | DPOINTS AND COVARIATES | 16 |
| | 5.1<br>5.2<br>5.3 | PRIMARY ENDPOINT | 17 |
| 6 | HA | NDLING OF MISSING VALUES | 17 |
| 7 | STA | ATISTICAL METHODOLOGY AND STATISTICAL ANALYSES | 18 |
| | | STATISTICAL METHODS STATISTICAL ANALYSES ADDITIONAL EXPLORATORY ANALYSIS umary | 18<br>21<br>21 |
| | | istical analysis description | |
| 8 | | RENGTH AND LIMITATION OF THE RESEACRCH METHODS | |
| 9 | | T OF TABLES AND TABLE SHELLS | |
| 1( | | FERENCES | |
| 11 | API | PENDICES | |
| | 11.1 | ANNEX 1 (Table 2): Study Variables and Definitions | 32 |

# 1 LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| AE | Adverse Event |
| AEM | Adverse Event Monitoring |
| BMI | Body Mass Index |
| CDC | Center for disease Control and prevention |
| COVID-19 | Corona Virus Disease 2019 caused by SARS-CoV-2 |
| eCRF | electronic Case Report Form |
| ECMO | extracorporeal mechanical oxygenation |
| EDC | Electronic Data Capture |
| EPIC-HR | Evaluation of Protease Inhibition for COVID-<br>19 in High-Risk Patients |
| ER | Emergency Room |
| EU | European Union |
| EUA | Emergency Use Authorization |
| FDA | Food and Drug Administration |
| GPP | Good Pharmacoepidemiology Practice |
| HCRU | Healthcare Resource Use |
| HFNC | High-flow nasal cannula |
| ICU | Intensive Care Unit |
| IEC | Independent Ethics Committee |
| IMV | Invasive Mechanical Ventilation |
| IRB | Institutional Review Board |

| Abbreviation | Definition |
|---|---|
| ISMF | Investigator Site Master File |
| KSA | Kingdom of Saudi Arabia |
| LOS | Length of Stay |
| MENA | Middle East and North Africa |
| NIH | National Institutes of Health |
| NIMV | Non-invasive Mechanical Ventilation |
| NIS | Non-interventional Study |
| NIV | Non Invasive Ventilation |
| PCR | Polymerase Chain Reaction |
| RWE | Real World Evidence |
| SAP | Statistical Analysis Plan |
| SAS | Statistical Analyses System |
| SARS-CoV-2 | Severe Acute Respiratory Syndrome<br>Coronavirus 2 |
| SOP | Standard Operating Procedure |
| STROBE | Strengthening the Reporting of Observational Studies in Epidemiology |
| USA | United States of America |
| PHEIC | Public Health Emergency of International<br>Concern |
| PhD | Doctor of Philosopy |
| WHO | World Health Organization |

# 2 AMENDMENTS FROM PREVIOUS VERSION(S)

| Version | <b>Effective Date</b> | <b>Change Type</b> | Section | <b>Summary of Revisions</b> |
|---|---|---|---|---|
| 1.0 | 22-May-2023 | Not Applicable | - | First version of SAP |
| 1.1 | 26-June-2023 | Amended | 7.2 Statistical<br>Analysis | Entire analysis content<br>for "Overall" only and<br>not stratified by Cohorts |
| | | Removed | 4.2 Subgroups | Section "Nirmatrelvir, ritonavir treatment completion (if available)" as data is not captured |
| | | New | 4.2 Subgroups | Days from COVID 19 symptoms onset to dispensing (if available) |
| | | New | 4.2 Subgroups | Days from COVID 19<br>symptoms onset to<br>nirmatrelvir, ritonavir<br>prescription (if<br>available) |
| | | Amended | 9 List of Tables and Table shells | Title of tables |
| 1.2 | 26-July-2023 | Amended | 3.1 Study Design | Updated patients section method |
| 1.3 | 16-August-2023 | Added | 4.2 Subgroups | Added analysis for<br>number of previous<br>COVID-19 infection |
| 1.4 | 31-August-2023 | Amended | 4.2 Subgroups | Removed Pre-omicron period subgroup analysis. |
| 1.5 | 05-December-<br>2023 | Added | 4.2 Subgroups | Stratifications added for COVID-19 variant and Duration to COVID-19 negative result(s) |
| | | Added | 7.2 Statistical<br>Analysis | Added analysis section<br>for COVID-19 variant<br>and Duration to<br>COVID-19 negative<br>result(s) |

| 2.0 | 16-September-<br>2024 | Amended | 3.1 Study Design | Sample size updated |
|---|---|---|---|---|
| | | Amended | 7.3 Additional exploratory analysis | <ul> <li>Additional analyses:</li> <li>Stratified analysis of Paxlovid prescription at index by demographic and clinical characteristics</li> <li>Stratified analysis of HCRU (Healthcare Resource use) at index date by demographic and clinical characteristics.</li> <li>Examine the association between patients' hospitalization due to COVID-19 related reasons and Covariates*, using logistic regression model at the index date.</li> </ul> |
| | | Amended | 9. List of tables and Table shells | As per additional exploratory analyses, list of tables updated, and corresponding table shells added in the excel. The analysis already performed influenced amendment mentioned in the section 7.3 |

#### 3 INTRODUCTION

Note: in this document, any text taken directly from the non-interventional (NI) study protocol is *italicised*. The protocol version 1.0 dated on 17 March 2023 was used to develop the SAP.

# **Background**

Coronaviruses are a group of viruses of zoonotic origin, of which seven species have been identified thus far as infectious to humans. In December, 2019, clusters of patients with idiopathic pneumonia were identified in Wuhan, China, with clinical presentation including fever, cough, dyspnea, and chest discomfort. A novel coronavirus sequence was isolated from the cluster of patients, termed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), with the associated respiratory disease termed COVID-19. By January 30th, 2020, the World Health Organization (WHO) declared COVID-19 a Public Health Emergency of International Concern (PHEIC) due to rapid community transmission via respiratory droplets, leading to an exponential surge in the number of cases and severity, especially in a context where knowledge on this novel virus' epidemiology and potentiality was scarce. COVID-19 was declared as a pandemic on 11 March 2020, and as of February 2023, more than 679 million cases and 6.8 million deaths have been confirmed globally in 228 countries and territories.

COVID-19 clinical presentation and severity is vastly heterogenous, whereby patients may experience asymptomatic infection, mild illness, moderate illness, severe illness, or critical illness requiring hospitalization. Common symptoms include cough, fever, dyspnea, fatigue, sore throat, anosmia, and nausea. Critical illness is characterized by severe respiratory failure, systemic inflammatory response, septic shock, and multisystem dysfunction and failure, including the cardiovascular system, central nervous system, gastrointestinal system, renal system, and skin. Recent data related to COVID-19 symptom severity have revealed that approximately 80% of cases are mild-to-moderate, 15% are severe, and 5% are critical. Whilst the majority of cases are indeed asymptomatic or mild, COVID-19 patients who are hospitalized due to infection are at great risk of prolonged disease, complications, increased hospital length of stay (LOS), high morbidity and mortality. I1-15

Based on the most recent treatment guidelines put forth by the National Institutes of Health (NIH), management of non-hospitalized adults with acute COVID-19 infection includes supportive care (e.g., adequate hydration, rest, monitoring body temperature, and taking antipyretics and analgesics to reduce symptom severity), advice on reducing viral transmission, and advice on when to seek healthcare provision or in-person evaluation. Adults that do not require hospitalization or supplemental oxygen yet are at high-risk of disease progression to severe/critical illness (eg, patients with malignancies, neurological diseases, hypertension, diabetes mellitus, obesity, and immunocompromised conditions), may additionally receive antiviral therapy to reduce risk of progression, hospitalization, or death. Current COVID-19 antiviral therapeutic options, in order of preference, include ritonavir-boosted nirmatrelvir (Paxlovid<sup>TM</sup>) or remdesivir. To

*Molnupiravir may additionally be considered as an alternative therapeutic option only when the aforementioned are unavailable, infeasible, or clinically inappropriate to use.*<sup>17</sup>

The Saudi MoH Protocol for Patients Suspected of/Confirmed with COVID-19 Supportive care and antiviral treatment of suspected or confirmed COVID-19 infection (Version 3.7) September 29th, 2022 follows the same guidance described above.<sup>18</sup>

Nirmatrelvir, ritonavir is an antiviral therapy consisting of two active substances that reduce the ability of SARS-CoV-2 to multiply in the body, and thus prevent disease progression. The first active substance, nirmatrelvir (PF-07321332), works by blocking viral enzyme activity and subsequent multiplication. The second active substance, ritonavir, delays breakdown of nirmatrelvir; thus, maintains sufficient levels of nirmatrelvir in the body to allow it to continue its effect on reducing viral multiplication. Nirmatrelvir, ritonavir should be initiated after confirmed COVID-19 diagnosis and within 5 days of symptom onset; administered as 300 mg of nirmatrelvir (two 150 mg tablets) with 100 mg ritonavir (one 100 mg tablet) together, every 12 hours, for 5 days. Based on the guidelines put forth by the Center for Disease Control and Prevention (CDC), COVID-19 patients who are at high-risk of disease progression to severe COVID-19 include patients aged >50 years, those who are unvaccinated or incompletely vaccinated, in addition to specific underlying medical conditions including asthma, cancer, chronic lung diseases, chronic liver diseases, Diabetes mellitus, and Down's syndrome.

Nirmatrelvir, ritonavir EUA was based on data from an interim analysis of a Phase II-III randomized, double-blind, placebo-controlled clinical trial in non-hospitalized adult patients with a confirmed COVID-19 diagnosis, who were symptomatic, and had at least 1 risk factor for progression to severe disease. 22,23 Interim analysis results from this trial, titled "Evaluation of Protease Inhibition for COVID-19 in High-Risk Patients (EPIC-HR)" (NCT04960202), revealed 89% reduced risk of COVID-19-related hospitalization and 28-day mortality among the Paxlovid group compared to the placebo group. 23,24 A meta-analysis on the efficacy and safety of nirmatrelvir, ritonavir for COVID-19 treatment has additionally shown an Overall 78% reduction in COVID-19-related mortality and hospitalization.<sup>24</sup> Whilst the trial was conducted prior to the emergence of the SARS-CoV-2 omicron variants, recent studies in real-world settings have shown that nirmatrelvir, ritonavir is also effective against these variants. 25-27 Other COVID-19 antiviral therapies with reported risk reduction of hospitalization or death include remdesivir (87% reduced risk), <sup>28</sup> sotrovimab (85% reduced risk), <sup>29</sup> and molnupiravir (50% reduced risk). 30 Sotrovimab is no longer authorized to treat COVID-19 in any *United States of America (USA) region due to increases in the proportion of COVID-19* cases caused by the Omicron BA.2 sub-variant. 31 Bebtelovimab has also been authorized for emergency use, and available data from the BLAZE-4 clinical trial have revealed reduced viral load and improvement in symptoms, however, no clinical efficacy data of patients at risk of progressing to severe COVID-19 is available vet. 32 Since November 2022 bebtelovimab is not currently authorized for emergency use in the USA because it is not expected to neutralize Omicron subvariants BQ.1 and BQ.1.1.<sup>33</sup>

Real-world studies assessing nirmatrelvir, ritonavir effectiveness and health impact are limited, and there are no studies yet that assess patients' treatment patterns. A real-world study conducted in Israel among high-risk patients showed nirmatrelvir, ritonavir to be highly effective, and was significantly associated with reducing the rate of progression to severe COVID-19 and COVID-19-specific mortality. Another study conducted in Hong Kong to assess the effectiveness of molnupiravir and nirmatrelvir, ritonavir during the Omicron BA.2 variant of COVID-19 among patients initially not requiring oxygen therapy revealed shorter time to achieve lower viral load, lower risk of disease progression, reduced hospital LOS, and lower risk of all-cause mortality. In Shanghai, China, results from a study assessing nirmatrelvir, ritonavir among immunocompromised inpatients further revealed treatment effectiveness in terms of faster viral load clearance, and shorter time to viral elimination, with patients having better prognosis when treatment was initiated ≤5 days following COVID-19 diagnosis. Shanghais in the study in the study assessing covidence of the study and the study assessing nirmatrelvir, ritonavir among immunocompromised in the study assessing nirmatrelvir, and study assessing nirmatrelvir, ritonavir among immunocompromised in the study assessing nirmatrelvir, ritonavir among immuno

Several countries have incorporated nirmatrelvir, ritonavir within their national COVID-19 treatment protocols after regulatory body approval for emergency use, including the USA,<sup>8</sup> several countries in Europe including the United Kingdom,<sup>36</sup> and European Union (EU) countries including Italy, Germany, and Belgium,<sup>19,37</sup> and the Middle East and North Africa (MENA) region, including the KSA and Bahrain.<sup>18,38</sup> Moreover, it is expected that additional countries will adopt the use of nirmatrelvir, ritonavir within their protocol as it becomes more readily available, particularly considering near-future decentralization and generic production of nirmatrelvir, ritonavir across a larger number of countries, including low- and middle-income countries.<sup>39</sup>

# Rationale

The COVID-19 pandemic has exacerbated healthcare systems globally, with dire repercussions on patients, healthcare infrastructure, resources, and finances. <sup>40</sup> Although COVID-19 patient characteristics and disease course in healthcare settings have been described in the literature since the beginning of the pandemic in various regions including the USA, <sup>41,42</sup> EU, <sup>43-45</sup> and the MENA region; <sup>46-48</sup> there is limited data related to COVID-19 patient characteristics, treatment patterns, and HCRU identified in an outpatient setting, particularly in the MENA region. One study reported that among other factors such as age, male gender, and underlying medical conditions; being of Arab ethnicity was associated with increased risk of severe COVID-19 and related mortality. <sup>26</sup>

In KSA, nirmatrelvir, ritonavir has been approved and conditionally registered by the Saudi Food and Drug Authority (SFDA) for patients aged  $\geq 12$  years, weighing  $\geq 40$  kg with mild-to-moderate COVID-19 symptoms and at high-risk for progression to severe COVID-19 infection. The availability of antiviral therapies such as nirmatrelvir, ritonavir in an outpatient setting has the ability to reduce disease progression, hospitalization, and COVID-19-related mortality, when eligible patients are treated. With the current EU authorization and subsequent use of nirmatrelvir, ritonavir, there is a need to generate -RWE during this early EUA utilization phase to inform decision-making on national levels.

As such, this study aims to describe the baseline demographic, clinical characteristics, and HCRU of adult COVID-19 patients who have been prescribed nirmatrelvir, ritonavir treatment in KSA.

#### 3.1 STUDY DESIGN

This is a multi-center, retrospective observational study that will be conducted in KSA. The aim of this study is to capture data on the baseline demographic, clinical characteristics, and HCRU of adult COVID-19 patients who have been prescribed nirmatrelvir, ritonavir treatment.

An overview of the study design is depicted in Figure 1. The sample size for this study depends on the number of COVID-19 patients visiting the selected sites, in addition to nirmatrelvir, ritonavir prescription practices by the treating physician in line with local prescription guidelines in KSA. However, based on feasibility assessments, the minimum target sample size for the study is approximately 250 evaluable patients across 3 sites in KSA. The study will aim to meet this target sample size with a single Cohort of patients identified retrospectively prior to the date of site initiation (Cohort 1); however, if the target sample size is not met, then a second Cohort of patients will be initiated after the site initiation date (Cohort 2).

#### Cohort 1:

The study will involve collection of pre-defined, structured data retrospectively from medical records (electronic and/or paper if necessary) of patients who meet the study eligibility criteria (see <u>Section 3.1.2</u>) and who have been prescribed nirmatrelvir, ritonavir treatment within a 15-month lookback period from the date of site initiation (Cohort 1). The lookback period will span from 01 April 2022 to 30 June 2023. Data abstracted from patients' medical records will include patient demographics and clinical characteristics at index date (defined as the date of nirmatrelvir, ritonavir treatment prescribing), in addition to patients' HCRU during the 30-day period post-index date.

### Cohort 2:

If the minimum target sample size of 250 patients is not achieved from Cohort 1, then a second Cohort of patients (Cohort 2) will be initiated and will be included in the study until the target sample size is met. Cohort 2 patients are those who meet the eligibility criteria (see Section 3.1.2), and who have been prescribed nirmatrelvir, ritonavir treatment after the date of site initiation. As for patients in Cohort 1, the following data will be collected for patients in Cohort 2: demographics and clinical characteristics at index date, and HCRU during the 30day period post-index date.

Patients in Cohort 1 will be enrolled in the study in a consecutive manner from start of site initiation till lookback period until we reach desired sample size, in case the number of eligible patients is significantly larger than the sample size<sup>52-54</sup>. For Cohort 2, patients will be enrolled in the study in a consecutive manner from start of site initiation until we reach desired sample size. *An electronic Case Report Form (eCRF) will be available for* 

the selected sites to fill in for each patient included in Cohort 1 or Cohort 2. Patient data will be extracted from the medical records and entered into the eCRFs by trained site study personnel. Participation in this study is not intended to change the routine treatment patients receive, as determined by their prescribing physicians; all treatment decisions, type and timing of the disease monitoring are per routine clinical care, and at the discretion of the treating physician and patient.

Figure 1. Study Design



# 3.1.1 Study population

Data will be collected for all eligible adult COVID-19 patients who have been prescribed nirmatrelvir, ritonavir across 3 selected sites in KSA which are National Guard Hospital-Riyadh, King Faisal Specialist Hospital-Riyadh and King Faisal Specialist Hospital-Jeddah. These 3 healthcare centers are the largest COVID-19 care providers in KSA representing the majority of COVID-19 patients who have been prescribed nirmatrelvir, ritonavir at the national level. In addition, these three healthcare centers have the same guidelines for treatment and management of patients with COVID-19.

The selected sites with well-established clinical research infrastructures, are situated in the major cities of KSA, where COVID-19 patients are most prevalent. They provide medical attention to any COVID-19 patient and provide healthcare to complicated patients, including immunocompromised patients.

These facilities also maintain patient records and have access to electronic medical records for patient data retrieval.

The minimum target sample size is 250 patients. Patient eligibility will be assessed at patient index date. Patients in Cohort 1 will be identified during a 15-month lookback period prior to the date of site initiation, and patients in Cohort 2 will be identified

following the date of site initiation if the minimum target sample size for the study is not achieved from Cohort 1.

#### 3.1.2 Inclusion Criteria

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

- 1. Confirmed COVID-19 infection during the study observation period.
- 2.  $Age \ge 18$  years old.
- 3. Nirmatrelvir, ritonavir written prescription.

#### 3.1.3 Exclusion Criteria

There are no exclusion criteria for this study.

#### 3.1.4 Data source

This is an observational, non-interventional study (NIS) involving retrospective collection of data throughout the observation period, obtained from the source outlined below.

• Medical records of patients prescribed nirmatrelvir; ritonavir: The authorized physician or study investigator will record patient demographics, clinical characteristics, COVID-19 vaccination history, nirmatrelvir, ritonavir prescription data, and HCRU data from patients' medical records into an eCRF.

All data collected in this study are intended to capture COVID-19 patient demographics, clinical characteristics, and patients' HCRU in a real-world setting. An eCRF will primarily be used for data collection, located on a secure web-based electronic data capture (EDC) system. The use of a standardised eCRF will ensure data is captured consistently across all sites. The eCRF must be signed by the investigator, and the signature serves to attest that the information contained in the eCRF is true. At all times, the investigator has the final responsibility for the accuracy and authenticity of all clinical and laboratory data entered into the eCRFs.

*Table 1 below depicts the data collection schedule for the study.* 

Table 1. Data Collection Schedule

| Variables | Cohort 1 | | Cohort 2 | |
|---|---|---|---|---|
| | Index date <sup>a</sup> | During the 30-day post-index period <sup>b</sup> | Index date <sup>a</sup> | During the 30-day post-index period <sup>c</sup> |
| Patient demographics | X | | X | |
| Patient clinical | X | | X | |
| characteristics | | | | |
| COVID-19 vaccination | X | | X | |
| history | | | | |
| COVID-19 infection data | X | X | X | X |
| Nirmatrelvir, ritonavir | X | | X | |
| prescription data | | | | |
| HCRU data | X | X | X | X |

COVID-19: Corona Virus Disease 2019 caused by SARS-CoV-2; HCRU: Healthcare Resource Use.

#### 3.1.5 Patient Medical Records

The authorized physician or study investigator will record patient demographics, clinical characteristics, COVID-19 vaccination history, nirmatrelvir, ritonavir prescription data, and HCRU data from patients' medical records into an eCRF.

# 3.2 STUDY OBJECTIVES

The aim of this study is to describe the baseline demographic, clinical characteristics, and HCRU of adult ( $\geq$ 18 years) COVID-19 patients who have been prescribed nirmatrelvir, ritonavir treatment.

# 3.2.1 Primary objective:

To describe the baseline demographic and clinical characteristics, including preexisting comorbidities, of adult COVID-19 patients who have been prescribed nirmatrelvir, ritonavir treatment.

## 3.2.2 Secondary objective:

To assess adult COVID-19 patients' HCRU within the 30-day period following nirmatrelvir, ritonavir prescription, including:

• Overall HCRU in inpatient and outpatient settings.

<sup>&</sup>lt;sup>a</sup> Cohort 1/Cohort 2: Index date is defined as the date of nirmatrelvir, ritonavir prescription.

<sup>&</sup>lt;sup>b</sup> Cohort 1: Post-index period is defined as the 30-day period after the index date and prior to the site initiation date.

 $<sup>^{</sup>c}$  Cohort 2: Post-index period is defined as the 30-day period after the index date and after the site initiation date.

#### 4 ANALYSIS SETS/POPULATIONS

#### 4.1 FULL ANALYSIS SET

The Full Analysis Set will contain all patient's data who fulfil the eligibility criteria (see Section 2.1.2).

#### 4.2 SUBGROUPS

Exploratory stratifications will be conducted, as appropriate and where the sample size permits, to explore differences by:

- Age groups: 18-49, 50-64, 65-74,  $\geq 75$  years of age;
- Gender:
- BMI categories:  $(<18.5 = underweight, 18.5-24.9 = normal, 25-29.9 = overweight, \ge 30 = obese)$ ;
- Smoking status;
- *Medications used to treat COVID-19 in addition to nirmatrelvir, ritonavir;*
- Previous COVID-19 infection;
- COVID-19 vaccination history;
- Nirmatrelvir, ritonavir treatment completion (if available)
- Days from COVID-19 diagnosis to nirmatrelvir, ritonavir index date;
- Days from prescription to dispensing (if available).
- Days from COVID 19 symptoms onset to dispensing (if available).
- Days from COVID 19 symptoms onset to nirmatrelvir, ritonavir prescription (if available).

For each stratification variable, the full analysis set will be segmented into non-overlapping subgroups based on the stratification variable values. The stratifications may not be meaningful, if there are no patient's data in some of the groups or there are many variables with a lot of missing data.

The exploratory stratifications will be conducted for the following study objectives if enough data are available:

Secondary objective: To assess adult COVID-19 patients' HCRU within the 30-day period following nirmatrelvir, ritonavir prescription, including: Overall HCRU in inpatient and outpatient settings.

The specific stratifications, and their corresponding reporting labels will be the following:

• Age groups: Age at time of PAXLOVID<sup>™</sup> prescription will be further categorized into 18–49, 50–64, 65–74, ≥75 years. Descriptive summary tables for subgroup analysis by defined age groups for the specified study objectives will be created as shown in *Table Shells 10*.

Gender (Male, Female); Descriptive summary tables for subgroup analysis by gender for the specified study objectives will be created as shown in **Table Shells** 11

- *BMI categories:* Body Mass Index (BMI) at time of PAXLOVID<sup>TM</sup> prescription will be further categorized as <18.5 = underweight, 18.5–24.9 = normal, 25–29.9 = overweight, ≥30 = obese. Descriptive summary tables for subgroup analysis by defined BMI categorization for the specified study objectives will be reported as shown in *Table Shells 12*.
- *Smoking status* (Never smoker; Former smoker; Current smoker); Descriptive summary tables for subgroup analysis by smoking status in terms of never smoker, former smoker and current smoker for the specified study objectives will be reported as shown in *Table Shells 13*.
- Medications used to treat COVID-19 in addition to nirmatrelvir, ritonavir;
   Descriptive summary tables for subgroup analysis by Medications used to treat COVID-19 in addition to nirmatrelvir, ritonavir at time of PAXLOVID™ prescription for the specified study objectives will be reported as shown in *Table Shells 14*.
- *Previous COVID-19 infection (Yes, No);* Descriptive summary tables for subgroup analysis by Previous COVID-19 infection for the specified study objectives will be created as shown in *Table Shells 15.* Additionally, Number of previous COVID-19 infections before the index date will be reported and further stratified by 0, 1, 2 and more. Descriptive summary tables for these groups will be reported as shown in *Table Shell 15.1* (If sufficient data available).
- *COVID-19 vaccination history;* Descriptive summary tables for subgroup analysis by COVID-19 vaccination history for the specified study objectives will be reported as shown in *Table Shells 16*.
- Days from COVID-19 diagnosis to nirmatrelvir, ritonavir index date; Duration in days from COVID-19 diagnosis to nirmatrelvir, ritonavir index date will be further categorized as 0-2 days, 3-5 days, more than/equal to 6 days. Descriptive summary tables for subgroup analysis by defined duration categorization for the specified study objectives will be reported as shown in *Table Shells 17*.
- Days from prescription to dispensing (if available): Duration in days from prescription to dispensing will be further categorized as 0-2 days, 3-5 days, more than/equal to 6 days. Descriptive summary tables for subgroup analysis by defined duration categorization for the specified study objectives will be reported as shown in Table Shells *Table Shells 18*.

- Days from COVID 19 symptoms onset to dispensing (if available): Duration in days from COVID 19 symptoms onset to dispensing as 0-2 days, 3-5 days, more than/equal to 6 days. Descriptive summary tables for subgroup analysis by defined duration categorization for the specified study objectives will be reported as shown in Table Shells *Table Shells 19*.
- Days from COVID 19 symptoms onset to nirmatrelvir, ritonavir prescription (if available): Duration in days from COVID 19 symptoms onset to prescription as 0-2 days, 3-5 days, more than/equal to 6 days. Descriptive summary tables for subgroup analysis by defined duration categorization for the specified study objectives will be reported as shown in Table Shells *Table Shells 20*.

Additionally, the exploratory stratifications will be conducted for COVID-19 variant and Duration to COVID-19 negative result(s) if enough data are available and will be reported as shown in Table Shells *Table Shells 22.1 to 22.7* and *Table Shells 23.1 to 23.10* respectively.

# 5 ENDPOINTS AND COVARIATES

Descriptive summary tabulations will describe the demographic, clinical characteristics as well as pre-existing comorbidities of the patients in the study population at the time of PAXLOVID<sup>TM</sup> prescription, and Healthcare Resource Use during the 30 days post index date.

#### 5.1 PRIMARY ENDPOINT

This study focuses on the patients who have received PAXLOVID<sup>TM</sup> for COVID-19 infection. The primary endpoints that describe the primary objectives in the study population will be:

- The baseline demographics (age, gender, ethnicity, education, employment status), clinical characteristics (height, weight, BMI, smoking status, pre-existing comorbidities), concomitant medications at index date and previous COVID-19 infection during the last 6 months, duration between last infection and index date, of the study population at the time of PAXLOVID<sup>TM</sup> prescription.
- COVID-19 vaccination history (Receipt of vaccination (yes/no), type of vaccine, duration between vaccination and Index date), number of doses, at the time of PAXLOVID<sup>TM</sup> prescription.
- Nirmatrelvir, Ritonavir prescription (total dose of Nirmatrelvir/Ritonavir, dose of Nirmatrelvir, dose of Ritonavir, Frequency of dose, dispensed amount) at the time of PAXLOVID<sup>TM</sup> prescription.

- Medications used to treat COVID-19 infection (Antiviral, Antiviral, Steroid, Antithrombotic, Monoclonal antibody, Hydroxychloroquine and Other medications) at the time of PAXLOVID<sup>TM</sup> prescription.
- HCRU characteristics in terms of patient hospitalization status, COVID-19 related hospitalization, length of days in the hospitalization due to COVID-19, Intensive care unit (ICU) admission and length of stay in the ICU due to COVID-19, supplemental oxygen use, vasopressor use, patient intubation, outpatient visits and ER Visits due to COVID-19 at the time of PAXLOVID™ prescription.

## 5.2 SECONDARY ENDPOINT

- HCRU characteristics in terms of patient hospitalization status, COVID-19 related hospitalization, length of days in the hospitalization due to COVID-19, Intensive care unit (ICU) admission and length of stay in the ICU due to COVID-19, supplemental oxygen use, vasopressor use, patient intubation, outpatient visits and ER Visits due to COVID-19 during the 30-day post-index period.
- COVID-19 PCR and/or antigen test result(s), PCR test result(s), Antigen test result (s), Duration to negative COVID-19 test during the 30 days post-index period.

## 5.3 COVARIATES AND VARIABLE DEFINITIONS

Table 2 depicts patient demographics, clinical characteristics, COVID-19 vaccination history, nirmatrelvir, ritonavir prescription data, COVID-19 infection, HCRU variables and Detailed operational definitions of variables.

Variables and detailed definitions of the variables are provided in <u>Table 2</u>.

# 6 HANDLING OF MISSING VALUES

Should missing data occur, the data will be analyzed as they are recorded in the eCRFs, and no imputation of missing data will be performed. The number of missing values for data elements will be reported.

All data analysis in this study will be performed on the Full Analysis Set containing all patients who fulfil the eligibility criteria, and thus missing data is not used as criteria for excluding the patients from the data analysis.

For both categorical and continuous variables, the amount of missing data will be reported. For categorical variables, the missing values will be analysed in the descriptive summary tables as a category. The missing values in the continuous variables will be ignored when calculating the summary statistics of mean, median, standard deviation, and quantiles.

If some of the variables of interest show to have a large amount or proportion of missing data, the summary statistics of the variable to be interpreted accordingly.

## 7 STATISTICAL METHODOLOGY AND STATISTICAL ANALYSES

## 7.1 STATISTICAL METHODS

This is a descriptive study, and as such, no statistical testing will be conducted. Analyses will be conducted using Statistical Analysis System (SAS) (version 9.3 or higher). Summary statistics for patient demographics, clinical characteristics, treatment patterns, and patient HCRU will be performed. Continuous variables will be summarized using standard summary statistics such as number of observations (n), mean, median, standard deviation (SD), first and third quartile, minimum and maximum value. Categorical variables will be summarized in frequency tables as counts and proportions of the total study population, and by subgroups where appropriate. The proportion of missing data will be reported for each variable.

Ad hoc population analyses would include stratification by demographic characteristics and presence of Underlying Medical Conditions Associated with Higher Risk for Severe COVID-19.

All patients who fulfill the study eligibility criteria will be included in the data set for analyses.

One interim analysis will be conducted after 3 months of recruitment only if the target sample size is not achieved from Cohort 1 i.e. Cohort 2 is initiated.

# 7.2 STATISTICAL ANALYSES

Note: Cohort 2 will be included in the study only if the target sample size is not achieved from Cohort 1.

Patients' enrollment will be summarized as shown in *Table Shell 1*.

Primary analysis: To describe the baseline demographic and clinical characteristics, including pre-existing comorbidities, of adult COVID-19 patients who have been prescribed nirmatrelvir, ritonavir treatment.

Patient and disease characteristics will be summarized using descriptive statistics. In terms of sociodemographic characteristics age, gender, ethnicity, education, and employment status will be reported as shown in *Table Shell 2*. Clinical characteristics in terms of weight, height, Body Mass Index (BMI), smoking status, pre-existing comorbidities, duration between pre-existing comorbidities and Index date in months, concomitant medications used to treat comorbidities at index date, most common concomitant medications (Trade name or generic name) for comorbidities, and most common Indication for comorbidities at index date will be reported as shown in *Table shell 3*.

Patient's COVID-19 vaccination history in terms of patient vaccinated/not vaccinated, total numbers of dose, type of vaccine, duration between vaccination and index date will be reported as shown in the *Table shell 4*.

Similarly, data on previous COVID-19 infection will be reported in terms of Number of previous COVID-19 infection, duration between previous infection to the index date, Medication used to treat previous COVID-19 infection as shown in the *Table shell 5*. COVID-19 Positive infection data at index date will be reported in terms of Type of COVID-19 Test (PCR or Antigen test), Result of COVID-19 Test (PCR or Antigen test), result of PCR test only, result of Antigen test only, duration between COVID-19 symptoms onset to index date, variant of COVID-19, medication used to treat the infection as shown in the *Table shell 6*.

Data related to Nirmatrelvir/Ritonavir prescription in terms of specialty of provider total dose of Nirmatrelvir/Ritonavir, in case of "other" dose specified of Nirmatrelvir and Ritonavir (if available), frequency, dispensed amount, type dispensed, days from COVID-19 diagnosis to nirmatrelvir, ritonavir at index date, days from prescription to dispensing (if available), days from COVID 19 symptoms onset to dispensing (if available) and days from COVID 19 symptoms onset to nirmatrelvir, ritonavir prescription (if available) will be summarized in descriptive statistics and reported as shown in the *Table shell 7*.

Data of Patient hospitalization, primary cause of patient hospitalization, length of hospitalization stay, Intensive Care Unit (ICU) admission, length of stay in Intensive Care Unit (ICU), supplemental oxygen use, type of oxygen, vasopressor use, patient intubation, outpatient visits, reason of outpatient visits, Emergency Room visits, and reason of Emergency Room visits at index date will reported as shown in the *Table shell* 8.

Secondary analysis: To assess adult COVID-19 patients' HCRU within the 30-day period following nirmatrelvir, ritonavir prescription, including: Overall HCRU in inpatient and outpatient settings.

Healthcare Resource Use (HCRU) data will be summarized using descriptive statistics in terms of patient hospitalization, number of time patient hospitalization, cause of patient hospitalization, length of stay in the hospitalization, Intensive Care Unit (ICU) admission,

number of Intensive Care Unit (ICU) admission, length of stay in Intensive Care Unit (ICU), supplemental oxygen use, type of oxygen, vasopressor use, patient intubation, outpatient visits, number of outpatient visits and reason of outpatient visits during the 30 days post index date and reported as shown in the *Table Shell 9*. Further stratification will be performed as described in <u>section 3.2</u>.

COVID-19 PCR and /antigen test result(s), Result(s) by PCR only, Result(s) by antigen test only, duration to COVID-19 negative result(s) by PCR and/antigen tests from the index date will be reported will be reported as shown in the *Table shell 21*.

COVID-19 variant by following stratifications will be reported as shown in the *Table shell 22.1 to 22.7:* (if sample size permits)

- Age groups: *Table shell 22.1*
- Gender: Table shell 22.2
- BMI categories: Table shell 22.3
- Smoking status: *Table shell 22.4*
- Previous COVID-19 infection: *Table shell 22.5*
- COVID-19 vaccination history: *Table shell 22.6*
- Underlying medical conditions: *Table shell 22.7*

Duration to COVID-19 negative result(s) by following stratifications will be reported as shown in the *Table shell 23.1 to 23.10:* (if sample size permits)

- Age groups: *Table shell 23.1*
- Gender: Table shell 23.2
- BMI categories: Table shell 23.3
- Smoking status: Table shell 23.4
- Previous COVID-19 infection: *Table shell 23.5*
- COVID-19 vaccination history: *Table shell 23.6*
- Underlying medical conditions: *Table shell 23.7*
- Medications used to treat COVID-19 in addition to nirmatrelvir, ritonavir: *Table shell 23.8*
- Days from COVID-19 diagnosis to nirmatrelvir, ritonavir index date: *Table shell* 23.9
- Days from prescription to dispensing (if available): **Table shell 23.10**

#### 7.3 ADDITIONAL EXPLORATORY ANALYSIS

# **Summary**

The following exploratory analysis will be conducted:

- 1. Stratified analysis of Paxlovid prescription at index by demographic and clinical characteristics.
- 2. Stratified analysis of HCRU (Healthcare Resource use) at index date by demographic and clinical characteristics.
- 3. Examine the association between patients' hospitalization due to COVID-19 related reasons at the index date and Covariates\*, using logistic regression model. \*Covariates: Age groups, Gender, BMI categories, smoking status, Pre-existing comorbidities, previous

# Statistical analysis description

1. "Stratified analysis of Paxlovid prescription at index by demographic and clinical characteristics"

Data related to Nirmatrelvir/Ritonavir prescription in terms of specialty of provider total dose of Nirmatrelvir/Ritonavir, in case of "other" dose specified of Nirmatrelvir and Ritonavir, frequency, dispensed amount, type dispensed, days from COVID-19 diagnosis to nirmatrelvir, ritonavir at index date, days from prescription to dispensing days from COVID-19 symptoms onset to dispensing and days from COVID-19 symptoms onset to nirmatrelvir, ritonavir prescription will be summarized in descriptive statistics by:

- Age groups: 18–49, 50–64, 65–74, >75 years
- Gender
- BMI categories: (<18.5 = underweight, 18.5-24.9 = normal, 25-29.9 = overweight,  $\ge 30$  = obese).
- Smoking status.
- Previous COVID-19 infection.
- COVID-19 vaccination history.

These tables will be reported as shown in the **table shells 7.1 to 7.6** 

2. "Stratified analysis of HCRU (Healthcare Resource use) at index date by demographic and clinical characteristics"

Data of Patient hospitalization, primary cause of patient hospitalization, length of hospitalization stay, Intensive Care Unit (ICU) admission, length of stay in Intensive Care Unit (ICU), supplemental oxygen use, type of oxygen, vasopressor use, patient intubation, outpatient visits, reason of outpatient visits, Emergency Room visits, and

reason of Emergency Room visits at index date will be summarized in descriptive statistics by:

- Age groups: 18-49, 50-64, 65-74,  $\ge 75$  years
- Gender
- BMI categories: (<18.5 = underweight, 18.5-24.9 = normal, 25-29.9 = overweight,  $\ge 30$  = obese).
- Smoking status.
- Previous COVID-19 infection.
- COVID-19 vaccination history.

  These tables will be reported as shown in the **table shells 8.1 to 8.6**.
- 3. "Examine the relationship between patients' hospitalization due to COVID-19 related reasons and various demographic and clinical factors at the index date."

We will be utilizing both univariate and multivariate binomial logistic regression to examine the association between patients' hospitalization due to COVID-19 at the index date and demographic and clinical factors mentioned below (covariates). All p-values will be reported as two-sided, and statistical significance will be determined at 0.05 alpha level. Separate univariate binary logistic regression model will be conducted for each covariate listed below and only covariates which will be found significant will be included in the Multivariate model along with clinically significant covariates (e.g BMI, Previous comorbidity status etc.). No interaction terms will be included in the model.

The following binary logistic regression equation will be used to model the relationship:

$$log(odds) = \beta_0 + \beta_1 X_1 + \beta_2 X_2 + ... + \beta_n * X_n$$

## Where:

- log(odds) represents the logarithm of the odds of the patients' hospitalization due to COVID-19
- $\beta_0$  is the intercept or constant term.
- $\beta_1$ ,  $\beta_2$ , ...,  $\beta_n$  are the coefficients associated with the independent variables (covariates)  $X_1$ ,  $X_2$ , ...,  $X_n$ .
- $X_1, X_2, ..., X_n$  are the values of the independent variables (Covariates)

Here,

**Outcome variable (Dependent variable):** patients' hospitalization due to COVID-19 related at index date (Yes=1/No\*\*=0).

\*\*No: No will include both "patients who had no hospitalization" as well as "patients with hospitalization due to non-COVID-19 related reasons".

# **Covariates (Independent variables):**

- Age groups (Reference group: 18-29 Year)
- Gender (Reference group: Female)
- BMI categories (Reference group: Normal)
- Smoking status (Reference group: Never smoke)
- Pre-existing comorbidities (Yes/No, Reference group: No)
- Previous COVID-19 infection (Yes/No, Reference group: No)
- COVID-19 vaccination history (Yes/No, Reference group: No)

The results will be presented in the terms of odd ratio (by exponentiating the logistic regression coefficient) and corresponding 95% CI. "p-values" and "confidence intervals (CIs)" will be obtained using statistical methods such as maximum likelihood estimation (MLE) or Wald tests.

These tables will be reported as shown in the table shells 24 to 24.1.

#### 8 STRENGTH AND LIMITATION OF THE RESEACRCH METHODS

# **Strengths**

The strength of this study includes use of patients' medical records for data collection, which allows data to be captured on a large, diverse cohort of patients with different characteristics in a quick and efficient manner.

Another strength is the eligibility criteria, which has been selected to be as broad as possible for the target patient population, so as to reflect the real-world clinical setting to the extent possible, and to minimize selection bias.

# **Limitations and Bias**

As this is a retrospective observational study and participant enrolment in the study will be done in a consecutive manner. This approach is associated with low possibility of bias and representativeness of the enrolled sample could be affected, if there is pattern observed among a particular age group or due to any season etc. In case such selection bias is observed, then additional stratification/ subgroup can be reported in the analysis, as required.

Since this study will involve collection of existing data from medical records, misclassification bias due to recording errors is possible. Medical records may not always be complete, the availability and quality/completeness of data may vary

considerably between different sites within KSA, and there may be abstraction errors and differences in reporting standards between the different sites.

Another limitation to be considered is the characteristics of the patient population to be included in the final analysis, which may potentially be biased based on the KSA national recommendations put in place for the management and treatment of COVID-19 during the observational period. This may affect the generalizability of findings from this study across different countries in the real-world setting.

At the patient-level, misclassification of drug exposure has to be considered. Medical records provide detailed information on patient demographics, clinical characteristics, and prescribed nirmatrelvir, ritonavir treatment, but may not contain information on the intended duration of use (days of supply) and may not contain accurate information on the actual treatment pattern of nirmatrelvir, ritonavir medications by the patient ie, patient adherence (if any).

COVID-19 outcomes are dependent on individuals seeking healthcare i.e., individual may have symptoms for long but if there is not an interaction with the health system, it will be unknown.

## 9 LIST OF TABLES AND TABLE SHELLS

| Number | Description |
|---|---|
| Table shells for Primary objectives | |
| Table shell 1 | Summary of patient enrolment at Index date. |
| Table shell 2 | Summary of demographic characteristics of patients at Index date. |
| Table shell 3 | Summary of clinical characteristics of patients at Index date. |
| Table shell 4 | Summary of COVID-19 vaccination history of patients at Index date. |
| Table shell 5 | Summary of previous COVID-19 infection of patients at Index date. |
| Table shell 6 | Summary of COVID-19 Positive infection of patients at Index date. |
| Table shell 7 | Summary of Nirmatrelvir/Ritonavir prescription at Index date. |
| Table shell 7.1 | Summary of Nirmatrelvir/Ritonavir prescription at index date by age groups. |
| Table shell 7.2 | Summary of Nirmatrelvir/Ritonavir prescription at index date by gender. |
| Table shell 7.3 | Summary of Nirmatrelvir/Ritonavir prescription at index date by BMI categories. |
| Table shell 7.4 | Summary of Nirmatrelvir/Ritonavir prescription at index date by smoking status. |
| Table shell 7.5 | Summary of Nirmatrelvir/Ritonavir prescription at index date by previous COVID-19 infection. |
| Table shell 7.6 | Summary of Nirmatrelvir/Ritonavir prescription at index date by COVID-19 vaccination history. |
| Table shell 8 | Summary of Healthcare Resource use at Index date. |

Table shell 21

| Table shell 8.1 | Summary of Healthcare Resource use at Index date by age groups. |
|---|---|
| Table shell 8.2 | Summary of Healthcare Resource use at index date by gender. |
| Table shell 8.3 | Summary of Healthcare Resource use at index date by BMI categories. |
| Table shell 8.4 | Summary of Healthcare Resource use at index date by smoking status. |
| Table shell 8.5 | Summary of Healthcare Resource use at index date by previous COVID-19 |
| | infection. |
| Table shell 8.6 | Summary of Healthcare Resource use at index date period by COVID-19 vaccination history. |

# Table shells for Secondary objectives

Table shell 9 Summary of Healthcare Resource use during the 30 days post index date period.

# Table shells for stratification analysis – Secondary objectives (HCRU)

| Table shells for s | difficultion unarysis Secondary objectives (Herke) |
|---|---|
| Table shell 10 | Summary of Healthcare Resource use during the 30 days post index date |
| | period by age groups. |
| Table shell 11 | Summary of Healthcare Resource use during the 30 days post index date |
| | period by gender. |
| Table shell 12 | Summary of Healthcare Resource use during the 30 days post index date |
| | period by BMI categories. |
| Table shell 13 | Summary of Healthcare Resource use during the 30 days post index date |
| | period by smoking status. |
| Table shell 14 | Summary of Healthcare Resource use during the 30 days post index date |
| | period by most common medication use to treat COVID-19 in addition to |
| | nirmatrelvir, ritonavir. |
| Table shell 15 | Summary of Healthcare Resource use during the 30 days post index date |
| | period by previous COVID-19 infection. |
| Table shell 15.1 | Summary of Healthcare Resource use during the 30 days post index date |
| | period by number of previous COVID-19 infection. |
| Table shell 16 | Summary of Healthcare Resource use during the 30 days post index date |
| | period by COVID-19 vaccination history. |
| Table shell 17 | Summary of Healthcare Resource use during the 30 days post index date |
| | period by days from COVID-19 diagnosis to nirmatrelvir, ritonavir |
| | prescription. |
| Table shell 18 | Summary of Healthcare Resource use during the 30 days post index date |
| | period by days from prescription to dispensing (if available). |
| Table shell 19 | Summary of Healthcare Resource use during the 30 days post index date |
| | period by days from COVID 19 symptoms onset to dispensing (if available). |
| Table shell 20 | Summary of Healthcare Resource use during the 30 days post index date |
| | period by days from COVID 19 symptoms onset to nirmatrelvir, ritonavir |
| | prescription (if available). |

post index date period. (If available)

Summary of COVID-19 PCR and /antigen test result(s) during the 30 days

| Table shell 22.1 | Summary of COVID-19 variant by age groups |
|---|---|
| Table shell 22.2 | Summary of COVID-19 variant by gender |
| Table shell 22.3 | Summary of COVID-19 variant by BMI categories |
| Table shell 22.4 | Summary of COVID-19 variant by smoking status |
| Table shell 22.5 | Summary of COVID-19 variant by previous COVID-19 infection |
| Table shell 22.6 | Summary of COVID-19 variant by COVID-19 vaccination history |
| Table shell 22.7 | Summary of COVID-19 variant by underlying medical conditions |
| Table shell 23.1 | Summary of duration to COVID-19 negative result(s) by age groups |
| Table shell 23.2 | Summary of duration to COVID-19 negative result(s) by gender |
| Table shell 23.3 | Summary of duration to COVID-19 negative result(s) by BMI categories |
| Table shell 23.4 | Summary of duration to COVID-19 negative result(s) by smoking status |
| Table shell 23.5 | Summary of duration to COVID-19 negative result(s) by previous COVID-19 infection |
| Table shell 23.6 | Summary of duration to COVID-19 negative result(s) by COVID-19 vaccination history |
| Table shell 23.7 | Summary of duration to COVID-19 negative result(s) by underlying medical conditions at index date |
| Table shell 23.8 | Summary of duration to COVID-19 negative result(s) by medications used to treat COVID-19 in addition to nirmatrelvir, ritonavir |
| Table shell 23.9 | Summary of duration to COVID-19 negative result(s) by days from COVID-19 diagnosis to nirmatrelvir, ritonavir index date |
| Table shell 23.10 | Summary of duration to COVID-19 negative result(s) by days from prescription to dispensing |
| Table shell 24 | Summary of patients' hospitalization due to COVID-19 related reasons at |
| | index date by covariates and univariate binary logistic models. |
| Table shell 24.1 | Summary of patients' hospitalization due to COVID-19 related reasons at |
| | index date by covariates and the <b>multivariable binary</b> logistic model |

## 10 REFERENCES

- 1. Hasöksüz M, Kiliç S, Saraç F. Coronaviruses and SARS-COV-2. Turk J Med Sci. 2020;50(Si-1):549-56.
- 2. Hu B, Guo H, Zhou P, Shi ZL. Characteristics of SARS-CoV-2 and COVID-19. Nat Rev Microbiol. 2021;19(3):141-54.
- 3. World Health Organization. COVID-19 Public Health Emergency of International Concern (PHEIC) Global research and innovation forum. 12 February 2020. [Available from: https://www.who.int/publications/m/item/covid-19-public-health-emergency-of-international-concern-(pheic)-global-research-and-innovation-forum] Accessed on October 11, 2022.

- 4. World Health Organization. WHO Situation Report 51 Coronavirus disease 2019 (COVID-19). 11 March 2020. [Available from: https://www.who.int/publications/m/item/situation-report---51] Accessed on October 11, 2022.
- 5. Worldometers. COVID Live- Coronavirus statistics. 11 October 2022. [Available from: https://www.worldometers.info/coronavirus/] Accessed on October 11, 2022.
- 6. Johns Hopkins Medicine. COVID Symptoms. 27 January 2022 [Available from: https://www.hopkinsmedicine.org/health/conditions-and-diseases/coronavirus/coronavirus-symptoms-frequently-asked-questions] Accessed on October 11, 2022.
- 7. Biancolella M, Colona VL, Mehrian-Shai R, Watt JL, Luzzatto L, Novelli G, et al. COVID-19 2022 update: transition of the pandemic to the endemic phase. Hum Genomics. 2022;16(1):19.
- 8. National Institutes of Health. Clinical Spectrum|COVID-19 Treatment Guidelines. 26 September 2022. [Available from: https://www.covid19treatmentguidelines.nih.gov/overview/clinical-spectrum/] Accessed on October 11, 2022.
- 9. Christiano D. Coronavirus symptoms: Mild, moderate, severe. 16 June 2022. [Available from: https://www.singlecare.com/blog/news/coronavirus-symptoms-and-incubation-period/] Accessed on October 11, 2022.
- 10. Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. Jama. 2020;323(13):1239-42.
- 11. Ginestra JC, Mitchell OJL, Anesi GL, Christie JD. COVID-19 Critical Illness: A Data-Driven Review. Annu Rev Med. 2022;73:95-111.
- 12. Tan E, Song J, Deane AM, Plummer MP. Global Impact of Coronavirus Disease 2019 Infection Requiring Admission to the ICU: A Systematic Review and Meta-analysis. Chest. 2021;159(2):524-36.
- 13. Domecq JP, Lal A, Sheldrick CR, Kumar VK, Boman K, Bolesta S, et al. Outcomes of Patients With Coronavirus Disease 2019 Receiving Organ Support Therapies: The International Viral Infection and Respiratory Illness Universal Study Registry. Crit Care Med. 2021;49(3):437-48.
- 14. Docherty AB, Harrison EM, Green CA, Hardwick HE, Pius R, Norman L, et al. Features of 20 133 UK patients in hospital with covid-19 using the ISARIC WHO

- Clinical Characterisation Protocol: prospective observational Cohort study. Bmj. 2020;369:m1985.
- 15. Richardson S, Hirsch JS, Narasimhan M, Crawford JM, McGinn T, Davidson KW, et al. Presenting Characteristics, Comorbidities, and Outcomes Among 5700 Patients Hospitalized With COVID-19 in the New York City Area. Jama. 2020;323(20):2052-9.
- 16. National Institutes of Health. Nonhospitalized Adults: General Management|COVID-19 Treatment Guidelines. 26 September 2022. [Available from: https://www.covid19treatmentguidelines.nih.gov/management/clinical-management-of-adults/nonhospitalized-adults-general-management/] Accessed on October 11, 2022.
- 17. National Institutes of Health. Nonhospitalized Adults: Therapeutic management|COVID-19 Treatment Guidelines. 26 September 2022. [Available from: https://www.covid19treatmentguidelines.nih.gov/tables/therapeutic-management-of-nonhospitalized-adults/] Accessed on October 11, 2022.
- 18. Saudi Ministry of Health. Saudi MoH Protocol for Patients Suspected of/Confirmed with COVID-19. 29 September 2022. [Available from: https://www.moh.gov.sa/Ministry/MediaCenter/Publications/Documents/MOH-therapeutic-protocol-for-COVID-19.pdf] Accessed on March 02, 2023.
- 19. European Medicines Agency. Paxlovid. 24 February 2022. [Available from: https://www.ema.europa.eu/en/medicines/human/EPAR/paxlovid] Accessed on October 11, 2022.
- 20. U.S. Food and Drug Administration. FDA Updates on Paxlovid for Health Care Providers. 4 May 2022. [Available from: https://www.fda.gov/drugs/news-events-human-drugs/fda-updates-paxlovid-health-care-providers] Accessed on October 11, 2022.
- 21. Centers for Disease Control and Prevention. Underlying medical conditions associated with higher risk for severe COVID-19: information for healthcare professionals. 5 December 2022. [Available from: https://www.cdc.gov/coronavirus/2019-ncov/hcp/clinical-care/underlyingconditions.html] Accessed on January 27, 2023.
- 22. Pfizer Inc. Pfizer announces additional phase 2/3 study results confirming robust efficacy of novel COVID-19 oral antiviral treatment candidate in reducing risk of hospitalization or death. 14 December 2021. [Available from: https://www.pfizer.com/news/press-release/press-release-detail/pfizer-announces-additional-phase-23-study-results] Accessed on October 11, 2022.

- 23. Mahase E. Covid-19: Pfizer's paxlovid is 89% effective in patients at risk of serious illness, company reports. BMJ. 2021;375:n2713.
- 24. Zheng Q, Ma P, Wang M, Cheng Y, Zhou M, Ye L, et al. Efficacy and safety of Paxlovid for COVID-19:a meta-analysis. J Infect. 2022.
- 25. Zhong W, Jiang X, Yang X, Feng T, Duan Z, Wang W, et al. The efficacy of paxlovid in elderly patients infected with SARS-CoV-2 omicron variants: Results of a non-randomized clinical trial. Front Med (Lausanne). 2022;9:980002.
- 26. Najjar-Debbiny R, Gronich N, Weber G, Khoury J, Amar M, Stein N, et al. Effectiveness of Paxlovid in Reducing Severe COVID-19 and Mortality in High Risk Patients. Clin Infect Dis. 2022.
- 27. Rai DK, Yurgelonis I, McMonagle P, Rothan HA, Hao L, Gribenko A, et al. Nirmatrelvir, an orally active Mpro inhibitor, is a potent inhibitor of SARS-CoV-2 Variants of Concern. bioRxiv. 2022:2022.01.17.476644.
- 28. Gottlieb RL, Vaca CE, Paredes R, Mera J, Webb BJ, Perez G, et al. Early Remdesivir to Prevent Progression to Severe Covid-19 in Outpatients. N Engl J Med. 2022;386(4):305-15.
- 29. Gupta A, Gonzalez-Rojas Y, Juarez E, Crespo Casal M, Moya J, Falci DR, et al. Early Treatment for Covid-19 with SARS-CoV-2 Neutralizing Antibody Sotrovimab. N Engl J Med. 2021;385(21):1941-50.
- 30. Mali KR, Eerike M, Raj GM, Bisoi D, Priyadarshini R, Ravi G, et al. Efficacy and safety of Molnupiravir in COVID-19 patients: a systematic review. Ir J Med Sci. 2022:1-14.
- 31. U.S. Food and Drug Administration. FDA updates sotrovimab emergency use authorization. 5 April 2022 [Available from: https://www.fda.gov/drugs/drugsafety-and-availability/fda-updates-sotrovimab-emergency-use-authorization] Accessed on October 11, 2022.
- 32. Lilly. Bebtelovimab|Emergency Use Authorization (EUA) for the Treatment of COVID-19 2022 [cited 2022. Available from: https://www.covid19.lilly.com/bebtelovimab.
- 33. U.S. Food and Drug Administration. FDA Announces bebtelovimab is not currently authorized in any US region [Available from: https://www.fda.gov/drugs/drugsafety-and-availability/fda-announces-bebtelovimab-not-currently-authorized-any-us-region] Accessed on October 11, 2022.
- 34. Wong CKH, Au ICH, Lau KTK, Lau EHY, Cowling BJ, Leung GM. Real-world effectiveness of molnupiravir and nirmatrelvir/ritonavir among COVID-19

- inpatients during Hong Kong's Omicron BA.2 wave: an observational study. medRxiv. 2022;2022.05.19.22275291.
- 35. Sun F, Lin Y, Wang X, Gao Y, Ye S. Paxlovid in patients who are immunocompromised and hospitalised with SARS-CoV-2 infection. The Lancet Infectious Diseases. 2022;22(9):1279.
- 36. National Institute for Health and Care Excellence. COVID-19 rapid guideline: Managing COVID-19. 10 July 2022 2022 [Available from: https://app.magicapp.org/#/guideline/L4Qb5n/section/EgaGN7] Accessed on October 11, 2022.
- 37. Italian Medicines Agency. Use of antivirals for COVID-19. February 2022. [Available from: https://aifa.gov.it/uso-degli-antivirali-orali-per-covid-19] Accessed on October 11, 2022.
- 38. Bahrain Ministry of Health. The Kingdom of Bahrain authorises the emergency use of oral COVID-19 antiviral, Paxlovid. 16 September 2022. [Available from: https://healthalert.gov.bh/en/article/News-627017] Accessed on October 11, 2022.
- 39. Pepperrell T, Ellis L, Wang J, Hill A. Barriers to Worldwide Access for Paxlovid, a New Treatment for COVID-19. Open Forum Infect Dis. 2022;9(9):ofac174.
- 40. Khetrapal S, Bhatia R. Impact of COVID-19 pandemic on health system & Sustainable Development Goal 3. Indian J Med Res. 2020;151(5):395-9.
- 41. Roth GA, Emmons-Bell S, Alger HM, Bradley SM, Das SR, de Lemos JA, et al. Trends in Patient Characteristics and COVID-19 In-Hospital Mortality in the United States During the COVID-19 Pandemic. JAMA Netw Open. 2021;4(5):e218828.
- 42. Peltan ID, Caldwell E, Admon AJ, Attia EF, Gundel SJ, Mathews KS, et al. Characteristics and Outcomes of US Patients Hospitalized With COVID-19. Am J Crit Care. 2022;31(2):146-57.
- 43. Giorgi Rossi P, Marino M, Formisano D, Venturelli F, Vicentini M, Grilli R. Characteristics and outcomes of a Cohort of COVID-19 patients in the Province of Reggio Emilia, Italy. PLoS One. 2020;15(8):e0238281.
- 44. Casas-Rojo JM, Antón-Santos JM, Millán-Núñez-Cortés J, Lumbreras-Bermejo C, Ramos-Rincón JM, Roy-Vallejo E, et al. Clinical characteristics of patients hospitalized with COVID-19 in Spain: Results from the SEMI-COVID-19 Registry. Rev Clin Esp (Barc). 2020;220(8):480-94.
- 45. Sjöström B, Månsson E, Viklund Kamienny J, Östberg E. Characteristics and definitive outcomes of COVID-19 patients admitted to a secondary hospital intensive care unit in Sweden. Health Sci Rep. 2021;4(4):e446.

- 46. Alharbi AA, Alqumaizi KI, Bin Hussain I, Alsabaani A, Arkoubi A, Alkaabba A, et al. Characteristics of Hospitalized COVID-19 Patients in the Four Southern Regions Under the Proposed Southern Business Unit of Saudi Arabia. Int J Gen Med. 2022;15:3573-82.
- 47. Araban M, Karimy M, Koohestani H, Montazeri A, Delaney D. Epidemiological and clinical characteristics of patients with COVID-19 in Islamic Republic of Iran. East Mediterr Health J. 2022;28(4):249-57.
- 48. Hassoun M, Alaywan L, Jaafouri H, Feghali R, Al-Mulki J, Radi F, et al. Clinical and epidemiological characteristics of the first 150 patients with COVID-19 in Lebanon: a prospective descriptive study. East Mediterr Health J. 2022;28(3):175-82.
- 49. von Elm E, Altman DG, Egger M, Pocock SJ, Gøtzsche PC, Vandenbroucke JP. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) Statement: guidelines for reporting observational studies. Int J Surg. 2014;12(12):1495-9.
- 50. International Committee of Medical Journal Editors (ICMJE). Recommendations for the Conduct, Reporting, Editing, and Publication of Scholarly Work in Medical Journals Updated May 2022 [Available from: https://www.icmje.org/icmje-recommendations.pdf.
- 51. WHO Working Group on the Clinical Characterisation and Management of COVID-19 infection. A minimal common outcome measure set for COVID-19 clinical research. Lancet Infect Dis.20(8):e192-e7.
- 52. BUJANG, M.A., 2017, Enhancement of systematic sampling for clinical survey: Systematic sampling with consecutive approach, Selangor: Institute of Graduate Studies, Universiti Teknologi Mara.
- 53. BOWERS, D., HOUSE, A. and OWENS, D., 2011, Carrying out a systematic search: Getting started in health research, United Kingdom: John Wiley and Sons Ltd
- 54. CHEW, B.H., SHARIFF-GHAZALI, S., MASTURA, I., HANIFF, J. and BUJANG, M.A., 2013, Age ≥ 60 years was an independent risk factor for diabetes-related complications despite good control of cardiovascular risk factors in patients with type2 diabetes mellitus, Exp Gerontol, 48(5):485–491. doi: 10.1016/j.exger.2013.02.017

# 11 APPENDICES

11.1 ANNEX 1 (TABLE 2): STUDY VARIABLES AND DEFINITIONS

| Variables | Role | Time point(s) | Operational definition |
|---|---|---|---|
| Age, Continuous | Patient demographics (Primary endpoint) | At index date | Age will be reported in year |
| Age, Category | Stratification variable | At index date | The age (Year) will be categorized as: • 18-49 Years • 50-64 Years • 65-74 Years • >75 Years |
| Gender | Patient demographics (Primary endpoint) | At index date | Gender (Sex) will be reported as: • Male • Female |
| Ethnicity | Patient<br>demographics<br>(Primary endpoint) | At index date | Ethnicity will be reported as: Arab Afro-Asian Asian/Pacific Islander Black/African American Hispanic/Latino Native American/Alaskan Native White/Caucasian, Multiracial/Biracial Unknown. Other [specify] |
| Education | Patient demographics (Primary endpoint) | At index date | Education will be reported as: No formal education Primary school Secondary school Undergraduate university degree Master's degree PhD or doctorate |
| Employment status | Patient demographics (Primary endpoint) | At index date | Employment status will be reported as: • Full-time employment • Part-time employment • Homemaker • Student • Retired • Disabled/too ill to work • Unemployed |

| Variables | Role | Time point(s) | Operational definition |
|---|---|---|---|
| Weight (kg) | Patient clinical characteristics (Primary endpoint) | At index date | Weight will be reported in kilograms (kg) |
| Height (m) | Patient clinical characteristics (Primary endpoint) | At index date | Height will be reported in meters (m) |
| BMI (kg/m²) | Patient clinical characteristics (Primary endpoint) | At index date | BMI will be calculated automatically based on the reported weight and height in the unit of kilograms over squared meters (kg/m²). |
| BMI category | Stratification variable | At index date | The calculated BMI will be categorized as: • Underweight (< 18.5) • Normal (18.5–24.9) • Overweight (25–29.9) • Obese (≥30) |
| Smoking Status | Patient clinical characteristics (Primary endpoint) | At index date | Smoking status will be reported as: Never smoker Former smoker Current smoker |
| Pre-existing comorbidities | Patient clinical characteristics (Primary endpoint) | At index date | Pre-existing comorbidities will be reported as: No Yes If yes, will be specified as: Diagnosis |
| Date of Pre-existing<br>Comorbidities onset | Patient clinical characteristics (Primary endpoint) | At index date | The date of onset of pre-existing comorbidities will be captured in (DD-MM-YYYY) |
| Duration between Pre-<br>existing comorbidities<br>onset to index date<br>(Months) | Patient clinical characteristics (Primary endpoint) | At index date | Duration between pre-existing comorbidities onset to index date will be calculated as: (Index date – Date of Pre-existing Comorbidities onset)/30.42 |
| Concomitant<br>medications for<br>comorbidities: Trade<br>name or generic name | Patient clinical characteristics (Primary endpoint) | At index date | Open field, all Concomitant medication will be reported. |
| Indication | Patient clinical characteristics (Primary endpoint) | At index date | Open field, all indication will be reported. |
| Date of initiation | Patient clinical characteristics (Primary endpoint) | At index date | The date of indication will be captured in (DD-MM-YYYY) |

| Variables | Role | Time point(s) | Operational definition |
|---|---|---|---|
| COVID-19 vaccination | COVID-19<br>vaccination history | At index date | History of COVID-19 vaccination will be reported as: • Yes • No |
| Number of COVID-19 vaccination dose | COVID-19<br>vaccination history | At index date | Number of doses will be calculated as: Total count of dose for each patient |
| Type of vaccination | COVID-19<br>vaccination history | At index date | Type of COVID-19 vaccination will be reported as: Protein-Serum Institute of India Protein-Novavax RNA-Moderna RNA-Pfizer/BioNTech Viral Vector-CanSino Viral Vector-Janssen Viral Vector-Janssen Viral Vector-Janssen Viral Vector-Janssen Inactivated-Serum Institute of India Inactivated-Bharat Biotech Inactivated-Sinopharm Inactivated-Sinopace |
| Date of vaccination<br>(For each dose) | COVID-19<br>vaccination history | At index date | The date of vaccination will be captured in (DD-MM-YYYY) |
| Duration between<br>vaccination and index<br>date (Months)<br>(For each dose) | COVID-19<br>vaccination history | At index date | Duration between vaccination<br>and index date (Months) will be<br>calculated as:<br>(Index date – Date of COVID-19<br>vaccination) /30.42 |
| Previous COVID-19 infection during the last 6 months | Previous COVID-19 infection | At index date | COVID-19 infection during last 6 month will be reported as: • Yes • No |
| Number of Previous<br>COVID-19 infection<br>during the last 6<br>months | Previous COVID-19 infection | At index date | Number of COVID-19 infection<br>during last 6 month will be<br>reported as count |
| Date of previous<br>COVID-19 infection<br>during the last 6 | Previous COVID-19 infection | At index date | Date of previous COVID-19 infection during the last 6 will be captured in (DD-MM-YYYY) |
| Duration between previous COVID-19 infection during the | Previous COVID-19 infection | At index date | Duration between previous<br>COVID-19 infection during last<br>6 month from index date will be<br>calculated as: |

| VariablesRoleTime point(s)Operational definitionlast 6 months and index date(Index date – Date of previous COVID-19 infection) /30.4Medication used to treat previous COVID-19 infectionAt index dateMedications used to treat previous COVID-19 infection during the last 6 will be replast 6 | |
|---|---|
| index date Medication used to treat previous COVID-19 infection Previous COVID-19 At index date previous COVID-19 infection Medications used to treat previous COVID-19 infection In infection during the during the during the last 6 will be rep | |
| Medication used to treat previous COVID-19 at index date treat previous COVID-19 infection during the Previous COVID-19 At index date previous COVID-19 infection during the last 6 will be rep | _ |
| treat previous COVID-<br>19 infection during the previous COVID-19 infection during the last 6 will be rep | |
| 19 infection during the during the last 6 will be rep | |
| 19 infection during the during the last 6 will be rep | on |
| • Antiviral (Yes; No) | ) |
| If yes, | |
| o Remdesivi | ſ |
| o Other, spec | ify |
| Antibiotic (Yes; No. | - |
| If yes, | |
| o Specify | |
| Steroid (Yes; No) | |
| If yes, | |
| o Budesonide | 2 |
| o Dexametha | |
| o Prednisolo | |
| ednisone | |
| o Hydrocorti | sone |
| o Methylpred | |
| one Sodium | |
| succinate | |
| o Other, spec | ifv |
| • Anti-thrombotic (Y | |
| No) | <b>C</b> 5, |
| If yes, | |
| o Enoxaparir | 1 |
| o Heparin | • |
| o Other, spec | ifv |
| Monoclonal antibo | - |
| (Yes; No) | ау |
| If yes, | |
| o Tocilizuma | h |
| o Other, spec | |
| Hydroxychloroquir | - |
| (Yes; No) | |
| If yes, | |
| o Specify | |
| Immunosuppressan | t |
| (Yes, No) | |
| If yes, | |
| o Baricitinib | ) |
| o Other, spec | |
| Intravenous immur | - |
| globulin (Yes, No) | |

| Variables | Role | Time point(s) | Operational definition |
|---|---|---|---|
| variables | Koic | Time point(s) | If yes, |
| | | | o Specify |
| | | | • Other medications (Yes; |
| | | | No) |
| | | | If yes, |
| | | | o Specify |
| Date of Positive | COVID-19 infection | At index date | Date of Positive COVID-19 |
| COVID-19 | data | | PCR/antigen test will be |
| PCR/antigen test | | | captured in (DD-MM-YYYY) |
| Date of COVID-19 | COVID-19 infection | At index date | Date of COVID-19 symptoms |
| symptoms onset | data | | onset will be captured in (DD- |
| | | | MM-YYYY) |
| Duration between | COVID-19 infection | At index date | Duration of COVID-19 |
| COVID-19 symptoms | data | | symptoms onset will be |
| onset and index date | data | | calculated as: |
| (Days) | | | (Index date – Date of COVID-19 |
| (Days) | | | symptoms onset) |
| COVID-19 variant | COVID-19 infection | At index date | Variant of COVID-19 will be |
| | | At index date | |
| (If available) | data | | reported as (if available): |
| | | | • Alpha [B.1.7 and Q] |
| | | | • Beta [B.1.351] |
| | | | • Gamma [P.1] |
| | | | • Delta [B.1.617.2; AY] |
| | | | • Epsilon [B.1.427; |
| | | | B.1.429] |
| | | | _ |
| | | | • Eta [B.1.525] |
| | | | • Iota [B.1.526] |
| | | | • Kappa |
| | | | [B.1.617.1];B.1.617.3; |
| | | | • Omicron [B.1.1.529; |
| | | | BA.1; BA.1.1; BA.2; |
| | | | BA.3; BA.4; BA.5] |
| | | | • Zeta [P.2] |
| | | | • Mu [B.1.621;B.1.621.1] |
| | | | • Omicron XBB.1.5. |
| 36.42 | COLUD 10 | 4.1.1.1. | • other [specify] |
| Medication use to treat | COVID-19 | At index date | Medications used to treat |
| COVID-19 infection | Medication data | | COVID-19 infection will be |
| | | | reported as: |
| | | | <ul> <li>Antiviral (Yes; No)</li> </ul> |
| | | | If yes, |
| | | | o Ritonavir |
| | | | <ul> <li>Other, specify</li> </ul> |
| | | | Antibiotic (Yes; No) |
| | | | If yes, |
| | | | o Specify |
| | | | <u> </u> |
| | | | <ul><li>Steroid (Yes; No)</li></ul> |

| Variables | Role | Time point(s) | Operational definition |
|---|---|---|---|
| | | | If yes, |
| | | | <ul> <li>Budesonide</li> </ul> |
| | | | <ul> <li>Dexamethasone</li> </ul> |
| | | | o Prednisolone/Pr |
| | | | ednisone |
| | | | <ul> <li>Hydrocortisone</li> </ul> |
| | | | <ul> <li>Methylprednisol</li> </ul> |
| | | | one Sodium |
| | | | succinate |
| | | | <ul> <li>Other, specify</li> </ul> |
| | | | <ul> <li>Anti-thrombotic (Yes;</li> </ul> |
| | | | No) |
| | | | If yes, |
| | | | <ul> <li>Enoxaparin</li> </ul> |
| | | | o Heparin |
| | | | o Other, specify |
| | | | <ul> <li>Monoclonal antibody</li> </ul> |
| | | | (Yes; No) |
| | | | If yes, |
| | | | <ul> <li>Infliximab</li> </ul> |
| | | | <ul> <li>Tocilizumab</li> </ul> |
| | | | <ul> <li>Other, specify</li> </ul> |
| | | | <ul> <li>Hydroxychloroquine</li> </ul> |
| | | | (Yes; No) |
| | | | If yes, |
| | | | o Specify |
| | | | <ul> <li>Immunosuppressant</li> </ul> |
| | | | (Yes, No) |
| | | | If yes, |
| | | | o Baricitinib |
| | | | <ul> <li>Other, specify</li> </ul> |
| | | | <ul> <li>Intravenous immune</li> </ul> |
| | | | globulin (Yes, No) |
| | | | If yes, |
| | | | o Specify |
| | | | • Other medications (Yes; |
| | | | No) |
| | | | If yes, |
| | | | o Specify |
| Prescription date | Nirmatrelvir, | At index date | Date of prescription of |
| (Index date) | ritonavir prescription | | Nirmatrelvir and Ritonavir will |
| | data | | be captured in (DD-MM-YYYY) |
| Specialty of provider | Nirmatrelvir, | At index date | Specialty of provider will be |
| | ritonavir prescription | | summarized as: |
| | data | | <ul> <li>Infectious Disease</li> </ul> |
| | | | <ul> <li>Internist</li> </ul> |
| | | | General Practitioner |

| Variables | Role | Time point(s) | Operational definition |
|---|---|---|---|
| | | | <ul> <li>Primary Care Physician</li> <li>ER</li> <li>Pulmonologist</li> <li>Other, specify</li> </ul> |
| Dose | Nirmatrelvir,<br>ritonavir prescription<br>data | At index date | Dose of Nirmatrelvir/Ritonavir will be reported as: • 300 mg (2x150)/100 mg • Other If Other, ○ Dose of Nirmatrelvir (Open field) ○ Dose of Ritonavir (Open field) |
| Frequency | Nirmatrelvir,<br>ritonavir prescription<br>data | At index date | Frequency of Nirmatrelvir/Ritonavir will be reported as: Twice a day Other If Other, Specify (Open field) |
| Dispensed amount | Nirmatrelvir,<br>ritonavir prescription<br>data | At index date | Open field: Will be captured by Box, Blister and Tablets. |
| Dispensed date (if available) | Nirmatrelvir,<br>ritonavir prescription<br>data | At index date | Date of dispensed will be captured in (DD-MM-YYYY) |
| Days from COVID-19<br>diagnosis to<br>nirmatrelvir, ritonavir<br>prescription date | Nirmatrelvir,<br>ritonavir prescription<br>data | At index date | Days from COVID-19 diagnosis to nirmatrelvir, ritonavir index date will be calculated as: [Prescription date (Index date)-Date of COVID-19 diagnosis] |
| Days from COVID-19<br>diagnosis to<br>nirmatrelvir, ritonavir<br>prescription date<br>(Categories) | Nirmatrelvir,<br>ritonavir prescription<br>data | At index date | Days from COVID-19 diagnosis to nirmatrelvir, ritonavir index date will be categorized as: • 0-2 days • 3-5 days • ≥ 6 days |
| Days from prescription to dispensing | Nirmatrelvir,<br>ritonavir prescription<br>data | At index date | Days from prescription to dispensing will be calculated as: [Dispensed date- Prescription date (Index date)] |
| Days from prescription<br>to dispensing<br>(Categories) | Nirmatrelvir,<br>ritonavir prescription<br>data | At index date | Days from prescription to dispensing will be categorized as: • 0-2 days • 3-5 days |

| Variables | Role | Time point(s) | Operational definition |
|---|---|---|---|
| | | | • ≥ 6 days |
| Days from COVID 19<br>symptoms onset to<br>dispensing (if<br>available) | Nirmatrelvir,<br>ritonavir prescription<br>data | At index date | Days from COVID 19 symptoms onset to dispensing will be calculated as: [Dispensed date- COVID-19 symptoms onset date] |
| Days from COVID 19<br>symptoms onset to<br>dispensing<br>(Categories) | Nirmatrelvir,<br>ritonavir prescription<br>data | At index date | Days from COVID 19 symptoms onset to dispensing will be categorized as: • 0-2 days • 3-5 days • ≥ 6 days |
| Days from COVID 19<br>symptoms onset to<br>nirmatrelvir, ritonavir<br>prescription (if<br>available) | Nirmatrelvir,<br>ritonavir prescription<br>data | At index date | Days from COVID 19 symptoms onset to nirmatrelvir, ritonavir prescription will be calculated as: [Prescription date (Index date) COVID-19 symptoms onset date] |
| Days from COVID 19<br>symptoms onset to<br>nirmatrelvir, ritonavir<br>prescription<br>(Categories) | Nirmatrelvir,<br>ritonavir prescription<br>data | At index date | Days from COVID 19 symptoms onset to nirmatrelvir, ritonavir prescription will be categorized as: • 0-2 days • 3-5 days • ≥ 6 days |
| Patient hospitalization | HCRU data | At index date | Patient hospitalization will be reported as: • Yes • No |
| Cause<br>(Patient<br>hospitalization) | HCRU data | At index date | Cause of patient hospitalization will be reported as (if available); • COVID-19 related • Non COVID-19 related |
| Outpatient setting | HCRU data | At index date | Outpatient setting will be defined if answer "No" to question "Patients hospitalization" |
| Length of Stay (Days) (Patient hospitalization) | HCRU data | At index date | Length of patients stay in hospitalization will be captured in days |
| Intensive Care Unit (ICU) admission | HCRU data | At index date | Intensive Care Unit (ICU) admission will be reported as: • Yes • No |

| Variables | Role | Time point(s) | Operational definition |
|---|---|---|---|
| Length of Stay (Days)<br>(ICU) | HCRU data | At index date | Length of patients in Intensive<br>Care Unit (ICU) will be captured<br>in days |
| Supplemental oxygen | HCRU data | At index date | Use of supplemental oxygen will be reported as: • Yes • No |
| Type of Supplemental oxygen | HCRU data | At index date | Type of supplemental oxygen use will be reported as: Oxygen mask Nasal prongs NIMV HFNC IMV ECMO |
| Vasopressor use | HCRU data | At index date | Use of Vasopressor will be reported as: Yes No |
| Patient intubation | HCRU data | At index date | Patient intubation data be reported as: • Yes • No |
| Outpatient visits | HCRU data | At index date | Outpatient visits data be reported as: • Yes • No |
| Cause (Outpatient visits) | HCRU data | At index date | Cause of Outpatient visits will be reported as (if available). • COVID-19 related • Non COVID-19 related |
| ER Visits | HCRU data | At index date | ER visits data be reported as: • Yes • No |
| Reason<br>(ER Visits) | HCRU data | At index date | Reason of ER visits will be reported as (if available); • COVID-19 related • Non COVID-19 related |
| Patient hospitalization | HCRU data | During the 30 day of post-index period | Patient hospitalization will be reported as: • Yes • No |
| Primary cause<br>(Patient<br>hospitalization) | HCRU data | During the 30 day of post-index period | Cause of patient hospitalization will be reported as (if available); • COVID-19 related • Non COVID-19 related |

| Variables | Role | Time point(s) | Operational definition |
|---|---|---|---|
| Outpatient setting | HCRU data | At index date | Outpatient setting will be |
| | | | defined if answer "No" to |
| | | | question "Patients |
| | | | hospitalization" |
| Length of Stay (Days) | HCRU data | During the 30 | Length of patients stay in |
| (Patient | | day of post- | hospitalization will be captured |
| hospitalization) | | index period | in days |
| Intensive Care Unit | HCRU data | During the 30 | Intensive Care Unit (ICU) |
| (ICU) admission | | day of post- | admission will be reported as: |
| | | index period | • Yes |
| | | | • No |
| Length of Stay (Days) | HCRU data | During the 30 | Length of patients in Intensive |
| (ICU) | | day of post- | Care Unit (ICU) will be captured |
| | | index period | in days |
| Supplemental oxygen | HCRU data | During the 30 | Use of supplemental oxygen will |
| | | day of post- | be reported as: |
| | | index period | • Yes |
| | | | • No |
| Type of Supplemental | HCRU data | During the 30 | Type of supplemental oxygen |
| oxygen | | day of post- | use will be reported as: |
| | | index period | Oxygen mask |
| | | F | Nasal prongs |
| | | | NIMV |
| | | | HFNC |
| | | | • IMV |
| | | | · · |
| Vasannasan | HCDH 1-4- | Description of the 20 | • ECMO |
| Vasopressor use | HCRU data | During the 30 | Use of Vasopressor will be |
| | | day of post- | reported as: |
| | | index period | • Yes |
| D. C. C. L. L. C. | HCDH 1 | D : 1 20 | • No |
| Patient intubation | HCRU data | During the 30 | Patient intubation data be |
| | | day of post- | reported as: |
| | | index period | • Yes |
| | | | • No |
| Outpatient visits | HCRU data | During the 30 | Outpatient visits data be reported |
| | | day of post- | as: |
| | | index period | • Yes |
| | | | • No |
| Cause | HCRU data | During the 30 | Cause of Outpatient visits will be |
| (Outpatient visits) | | day of post- | reported as (if available); |
| | | index period | <ul> <li>COVID-19 related</li> </ul> |
| | | | <ul> <li>Non COVID-19 related</li> </ul> |
| ER Visits | HCRU data | During the 30 | ER visits data be reported as: |
| | | day of post- | • Yes |
| | | index period | • No |

| Variables | Role | Time point(s) | Operational definition |
|---|---|---|---|
| Reason | HCRU data | During the 30 | Reason of ER visits will be |
| (ER Visits) | | day of post- | reported as (if available); |
| | | index period | COVID-19 related |
| | | | Non COVID-19 related |
| COVID-19 PCR and / | COVID-19 infection | During the 30 | COVID-19 PCR and / or antigen |
| or antigen test result(s) | data | day of post- | test result(s) will be reported as: |
| (If available) | uata | index period | <ul> <li>Positive</li> </ul> |
| | | | <ul> <li>Negative</li> </ul> |
| | | | Indeterminate |
| COVID-19 PCR result | COVID-19 infection | During the 30 | COVID-19 PCR test result will |
| (If available) | data | day of post- | be reported as: |
| | uata | index period | <ul> <li>Positive</li> </ul> |
| | | | <ul> <li>Negative</li> </ul> |
| | | | <ul> <li>Indeterminate</li> </ul> |
| COVID-19 Antigen | COVID-19 infection | During the 30 | COVID-19 Antigen test result |
| test result | data | day of post- | will be reported as: |
| (If available) | uata | index period | <ul> <li>Positive</li> </ul> |
| | | | <ul> <li>Negative</li> </ul> |
| | | | <ul> <li>Indeterminate</li> </ul> |
| Date of COVID-19 | COVID-19 infection | During the 30 | Date of COVID-19 PCR/antigen |
| PCR/antigen test | data | day of post- | test will be captured in (DD- |
| | uata | index period | MM-YYYY) |
| Duration to Negative | COVID-19 infection | During the 30 | Duration to negative COVID-19 |
| COVID-19 test | data | day of post- | test after initiation of |
| (Months) | uata | index period | Nirmatrelvir, Ritonavir will be |
| | | | calculated as: |
| | | | (Date of Negative COVID-19 |
| | | | result - Index date)/30.42 |

COVID-19: Corona Virus Disease 2019 caused by SARS-CoV-2; PhD: Doctor of Philosophy; BMI: body mass index; PCR: polymerase chain reaction; ECMO: extracorporeal mechanical oxygenation; ER: emergency room; HCRU: Healthcare Resource Use; HFNC: high-flow nasal cannula; IMV: invasive mechanical ventilation; LOS: length of stay; NIMV: non-invasive mechanical ventilation